CLINICAL TRIAL: NCT06294769
Title: Effect of Aromatherapy on Postoperative Pain in Adult Patients in Post-anesthesics Recovering Room: Randomized Clinical Trial
Brief Title: Effect of Aromatherapy on Postoperative Pain: Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Maria Fernanda de Oliveira Faria, Investigador Maria Fernanda, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 022024 Maria Fernanda
Record Dates: First submitted 2024-02-14; First posted 2024-03-06 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Acute Pain; Perioperative/Postoperative Complications; CAM; Nurse's Role
Keywords: Acute Pain; Perioperative Nursing; Aromatherapy
MeSH Terms: conditions — Acute Pain; Postoperative Complications

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: 2% lavender essential oil. (Experimental): Group will receive application of aromatherapy with 2% lavender essential oil dermal and inhalation via by a nurse, associated with usual care, in the immediate postoperative period.
  Interventions: Other: essencial oil of lavandula angustifolia
- Group 2: grape seed vegetable oil. (Placebo Comparator): Placebo group will only receive the application of grape seed vegetable oil associated with usual care in the post anesthetic recovery room.
  Interventions: Other: grape seed vegetable oil

INTERVENTIONS:
Other: essencial oil of lavandula angustifolia — The intervention will consist of the application of aromatherapy with 2% lavender essential oil cutaneously and inhalation via by a nurse, associated with usual care, in the immediate postoperative period
  Arms: Group 1: 2% lavender essential oil.
Other: grape seed vegetable oil — The placebo group will only receive the application of grape seed vegetable oil associated with usual care in the immediate postoperative period.
  Arms: Group 2: grape seed vegetable oil.

SUMMARY:
Introduction: Pain is one of the main complications in the immediate postoperative period that can harm the patient and can be managed through pharmacological and non-pharmacological methods. Complementary Integrative Health Practices are non-pharmacological methods that use therapeutic resources based on traditional knowledge to treat symptoms. Among them, aromatherapy stands out, which consists of the use of essential oils through inhalation or topical application for therapeutic purposes and which can be used as a nursing intervention, especially in the context of perioperative care. Objective: To evaluate the effect of aromatherapy on postoperative pain in adult patients in the immediate postoperative period. Method: This is a randomized controlled clinical trial that will be carried out in a teaching hospital. The project was submitted to the Research Ethics Committees of the School of Nursing of the University of Sao Paulo and the University of Sao Paulo Hospital. Adult patients undergoing elective surgical procedures of any surgical specialty under anesthesia of any type will be included. Individuals diagnosed with dementia, cognitive impairment or chronic pain will be excluded; individuals with a history of asthma, allergic bronchitis, chronic obstructive pulmonary disease, contact dermatitis or allergy to cosmetics with lavender fragrance, or hypersensitivity to the compounds used in the intervention; procedure for reoperation for any reason. The intervention will consist of the application of aromatherapy with 2% lavender essential oil through the skin and inhalation by a nurse, associated with usual care, in the immediate postoperative period; the placebo group will only receive the application of grape seed vegetable oil associated with usual care. A numerical verbal scale will be applied to assess pain and vital parameters will be measured upon patient admission, every fifteen minutes in the first hour and every thirty minutes in the second hour or after 15, 30, 45, 60 minutes, 1h30 minutes and 2 hours after applying the intervention, in the post-anesthesia recovery room. Possible associations between variables will be verified using Pearson's Chi-square or Fisher's exact tests. Comparison between means or medians will be made using the Student's t or Mann-Whitney tests, depending on the normality determined according to the Kolmogorov-Smirnov test. The significance level adopted will be 5%.

ELIGIBILITY:
Inclusion Criteria:

* adult patients undergoing elective surgical procedures of any surgical specialty under anesthesia of any type

Exclusion Criteria:

* individuals diagnosed with dementia, cognitive impairment or chronic pain;
* individuals with a history of asthma, allergic bronchitis, chronic obstructive pulmonary disease, contact dermatitis or allergy to cosmetics with lavender fragrance, or hypersensitivity to the compounds used in the intervention;
* procedure for reoperation for any reason

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 138 (Actual)
Dates: Start 2024-03-18 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Acute pain | 2 hours
  A numerical verbal scale (1 to 10) for assessing pain upon patient admission, after 15, 30, 45, 60 minutes, 1h30 minutes and 2 hours after application intervention, in the post-anesthesia recovery room.

SECONDARY OUTCOMES:
Blood pressure (both systolic and diastolic) | 2 hours
  Non-invasive blood pressure measurement (in mmHg) upon patient admission, after 15, 30, 45, 60 minutes, 1h30 minutes and 2 hours after application intervention, in the post-anesthesia recovery room
Heart rate | 2 hours
  Heart rate measurement with multi parameter monitor(in bpm) upon patient admission, after 15, 30, 45, 60 minutes, 1h30 minutes and 2 hours after application intervention, in the post-anesthesia recovery room
Respiratory frequency | 2 hours
  Respiratory frequency assessment (breathing rate by counting the number of breaths per minute) upon patient admission, after 15, 30, 45, 60 minutes, 1h30 minutes and 2 hours after application intervention, in the post-anesthesia recovery room
Oxygen saturation | 2 hours
  Oxygen saturation (SpO2) measurement (in percent (%), with a pulse oximeter non-invasive device) upon patient admission, after 15, 30, 45, 60 minutes, 1h30 minutes and 2 hours after application intervention, in the post-anesthesia recovery room
Temperature | 2 hours
  Temperature assessment (in Celsius scale ) upon patient admission, after 15, 30, 45, 60 minutes, 1h30 minutes and 2 hours after application intervention, in the post-anesthesia recovery room

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade de São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No